CLINICAL TRIAL: NCT04980703
Title: Grain Moxibustion Treatment on Insomnia: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYS20210601
Record Dates: First submitted 2021-06-28; First posted 2021-07-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: moxibustion; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grain moxibustion (Experimental): Grain moxibustion +standard care
  Interventions: Device: Grain moxibustion
- Sham grain moxibustion (Sham Comparator): Sham grain moxibustion +standard care
  Interventions: Device: Sham grain moxibustion
- Wait-list control (Other): Standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Grain moxibustion — Take Baihui(GV20), apply vaseline on the acupoint, knead moxa villi into grain size, put it on GV20, and ignite it with incense. When the patient feels burning or a little pain, put out moxa with gauze and keep for 10 seconds, so as to ensure enough heat to be penetrated into the acupoint. There are 3 cones for the first six times and 5 cones for the last six times . After the treatment of GV20, the patient will be in prone position. Select bilateral Xinshu(BL15) and Pishu(BL20) and operate the same as that of GV20. 3 times a week, 12 times in all. During the trial, patients with severe sleep disorders will be allowed to take the sedative-hypnotic drug eszopiclone 0.5-2mg orally (Sinopharm approval H31021534, Shanghai Shangyao Xinyi Pharmaceutical Co., Ltd.).
  Arms: Grain moxibustion
Device: Sham grain moxibustion — Take Baihui(GV20), apply vaseline on the acupoint, knead moxa villi into grain size, put it on GV20, and ignite it with incense. When the moxa burns to half （the patient hasn't feel hot or feel a little hot）, take the moxa away with tweezers. There are 3 cones for the first six times and 5 cones for the last six times . After the treatment of GV20, the patient will be in prone position. Select bilateral Xinshu(BL15) and Pishu(BL20) and operate the same as that of GV20. 3 times a week, 12 times in all. During the trial, patients with severe sleep disorders will be allowed to take the sedative-hypnotic drug eszopiclone 0.5-2mg orally (Sinopharm approval H31021534, Shanghai Shangyao Xinyi Pharmaceutical Co., Ltd.).
  Arms: Sham grain moxibustion
Other: Standard care — Participants in the wait-list control with severe sleep disorders will be allowed to take the sedative-hypnotic drug eszopiclone 0.5-2mg orally (Sinopharm approval H31021534, Shanghai Shangyao Xinyi Pharmaceutical Co., Ltd.). And after waiting for 12 weeks, these patients will be treated with the same grain moxibustion as the grain moxibustion group.
  Arms: Wait-list control

SUMMARY:
This trial intends to observe the clinical efficacy and safety of grain moxibustion at Baihui(GV20), Xinshu(BL15) and Pishu(BL20) in the treatment of insomnia.

DETAILED DESCRIPTION:
Insomnia is one of the most common sleep disorders. The main symptoms are difficulty in falling asleep, decreased sleep quality and sleep time, and affect the normal work, study and life during the day.

Acupuncture has a good clinical effect on insomnia, but most of the treatment methods are acupuncture or electroacupuncture. Moxibustion therapy, as one of the main components of the therapy, has the advantages of simple operation, wide acceptance, which is suitable for a wide range of promotion and application.At present, the trials of moxibustion in the treatment of insomnia mainly focus on mild moxibustion. The number of studies is small, and the research is designed insufficiently, so it is difficult to draw a positive conclusion, and needs to be further confirmed by rigorous designed experiments. In addition, grain moxibustion, which is widely used in clinic, has the advantages of more convenient operation, short treatment time and strong permeability. However, its efficacy and safety in the treatment of insomnia are still unclear, so it is necessary to carry out a randomized controlled trial to confirm it.

One hundred and two eligible patients will be randomly assigned to one of 3 groups: grain moxibustion group, sham grain moxibustion group and wait-list control group. Treatment will be given 3 times per week for 4 weeks. The primary outcome is the Pittsburgh Sleep Quality Index (PSQI). The secondary outcomes are changes of PSQI scores from baseline to 8 week follow-up, sleep monitoring of bracelet, Athens Insomnia Scale（AIS）, Generalized Anxiety Disorder Scale-7 (GAD-7), Patient Health Questionnaire-9 (PHQ-9) and recurrence observation during the follow-up period. Daily dose of patients' estazolam will be recorded in the dairy. All adverse effects will be assessed by the Treatment Emergent Symptom Scale (TESS). Outcomes will be evaluated at baseline, 4 weeks post-treatment, as well as at 8 week and 12 week follow-up.

This trial intends to observe the clinical efficacy and safety of grain moxibustion at Baihui(GV20), Xinshu(BL15) and Pishu(BL20) in the treatment of insomnia, which will provide an experimental basis for the treatment of insomnia with grain moxibustion and lay the foundation for the promotion and application of moxibustion in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of insomnia;
2. TCM syndrome differentiation belongs to deficiency of both heart and spleen;
3. Male or female participants aged 18-75;
4. Participants whose PSQI score is 5-15;
5. The course of disease is more than 3 months;
6. Participants who voluntarily agree with the investigation and sign a written informed consent form for the clinical trial.

Exclusion Criteria:

1. Participants with mental retardation;
2. Participants with serious cardiovascular diseases, liver, kidney and hematopoietic system diseases;
3. Insomnia is caused by nervous system diseases (such as stroke, Parkinson's disease) or mental disorders (including depression or anxiety);
4. Female participants who is pregnant or lactating;
5. Participants with diabetes and sensory dysfunction.
6. Participants with skin diseases of acupoints;
7. Taking sedative hypnotics (including barbiturates, benzodiazepines, tranquilizers, diphenylmethane, etc) and other insomnia related drugs within 2 weeks before the trial;
8. Participants with dependence on sleeping drugs;
9. Participants suffering from malignant tumor, sequelae of severe cerebral apoplexy, organ failure and other major diseases that affect insomnia and therapeutic effect.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2027-07-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Pittsburgh Sleep Quality Index (PSQI) | Baseline and week 4
  The Pittsburgh Sleep Quality Index (PSQI) is a widely-used questionnaire to assess one's sleep disorders over one month. It is comprised of 19 self-rated items and 5 other-rated items. The scores include the following indicators: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of medication, and daytime dysfunction. Each indicator is rated from 0 to 3. The accumulated scores of the seven indicators constitute the total score of PSQI (0-21). The higher score indicates the worse sleep quality and severer sleep disorders. The investigators set the changes of PSQI scores between baseline to week 4 as the primary outcome, to evaluate the effectiveness of acupuncture for depression related insomnia.

SECONDARY OUTCOMES:
Changes of PSQI scores | Baseline and week 12
  As is mentioned above, PSQI is a widely-used questionnaire to assess one's sleep disorders over one month. In order to assess the effects of acupuncture on patients' sleep quality during the intervention period, and to assess the durative effects of acupuncture after the intervention ends, the investigators set the changes of PSQI scores between baseline to week 8 and week 12 as the secondary outcome.
Sleep monitoring of bracelet | Week 12
  Xiaomi Bracelet 3(XMSH05HM)will be worn on the wrist of the participants, recording the sleep time at night, deep sleep time, light sleep time, awake time, time to fall asleep last night and time to wake up this morning.
Changes of Athens Insomnia Scale(AIS) | Baseline and week 12
  Using the Athens Insomnia Scale to test the subjective sleep quality of patients. It is comprised of 8 items. The range were from 0-3. Total score < 4 means sleep well; total score =4-6 means suspicious of insomnia; total score > 6 means insomnia. The changes of AIS scores between baseline to week 4, week 8 and week 12 are the secondary outcome.
Changes of Generalized Anxiety Disorder Scale-7(GAD-7) | Baseline and week 12
  Changes in anxiety will be measured using the Generalized Anxiety Disorder Scale (GAD-7), which contains 7 items with total scores ranging from 0 to 21. Scores of 5, 10, and 15 are cut-offs for mild, moderate, and severe anxiety, respectively. An add-on item assessing the patient's global impression of symptom-related impairment helps researchers understand the extent to which anxiety interferes in daily life. The GAD-7 has factorial validity for the diagnosis of general anxiety disorder and is sensitive to change. The changes of GAD-7 scores between baseline to week 4, week 8 and week 12 are the secondary outcome.
Changes of Patient Health Questionnaire-9 (PHQ-9) | Baseline and week 12
  Changes in depressive symptoms will be measured using the 9-item Patient Health Questionnaire-9 (PHQ-9) to assess depressive symptoms. With total scores ranging from 0 to 27, scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression, respectively. The PHQ-9 has factorial validity for the diagnosis of major depressive disorder. The changes of PHQ-9 scores between baseline to week 4, week 8 and week 12 are the secondary outcome.
Recurrence observation during the follow-up period | Week 12
  In case of relapse (PSQI score increase rate > 50% or need to adjust drugs to control the disease) or serious adverse reactions during the follow-up period, the time from the beginning to the end of treatment , the specific medication plan and the state of illness during the follow-up period will be recorded. The recurrence rate and average recurrence time during the follow-up period will be calculated according to the number of recurrence within week 4 to week 12 follow-up in each group.
Dose dairy | 12 weeks
  Compare the use rate and dosage of estazolam during treatment and follow-up.

OTHER OUTCOMES:
Blind evaluation | Week 4
  The participants will be asked to predict whether they were treated by grain moxibustion or sham grain moxibustion according to their self feelings.
Abnormalities after the moxibustion | Week 4
  Abnormalities after the moxibustion are skin scald, blistering or other discomfort caused by the moxibustion. Doctors will always have a burn ointment to prevent burns. If the patient gets a blister, the doctor will deal with it in time and inform the patient of the follow-up protective measures.

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, PhD, MD, Study Chair — Shanghai Institute of Acupuncture and Meridian
Locations (1):
- Shanghai Institute of Acupuncture, Moxibustion and Meridian, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be maintained by the principal investigator. Other investigators may consult with the principal investigator.
Supporting Information: Study Protocol
Time Frame: The protocol will be published online and is expected to be available in one to two years.
Access Criteria: Open up online for everyone.